CLINICAL TRIAL: NCT00822588
Title: A Prospective, Randomized, Controlled Trial of Retransfusion of Intra-operatively Collected Filtered Whole Blood in Total Hip Surgery
Brief Title: Comparison in Need for Bank Blood Between Patients Undergoing Total Hip Surgery That Either Receive Their Own Blood Back or Not
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YA-DRA-0001
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Arthroplasty, Replacement, Hip; Blood Transfusion; Blood Transfusion, Autologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Sangvia® System
- 2 (No Intervention)

INTERVENTIONS:
Device: Sangvia® System — Sangvia® Intra- and Post-op System
  Arms: 1

SUMMARY:
The study is a prospective, controlled, randomised and assessor blind study that investigate if the need for bank blood transfusion could be reduced in patients, undergoing primary or revision total hip replacement surgery, who receive their own blood back with the medical device Sangvia.

A comparison in need for bank blood will be made between patients that either receive their own blood back or not.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Scheduled for primary or secondary, cemented or non-cemented, total hip arthroplasty
* Classified as ASA Physical Status Classification System class P1, P2 or P3 according to the American Society of Anaesthesiology.

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study site)
* Previous enrollment or randomisation of treatment in the present study
* Expected or confirmed participation in another clinical study, that may interfere with the present study, during the study period
* Suspected severe non-compliance to protocol as judged by the investigator
* Current symptoms of haemophilia
* Current symptoms of hyperkalaemia
* Current symptoms of systemic infection or local infection in the operation field
* Current symptoms of impaired renal function including creatinine/clearance levels above the normal reference values
* History of or presence of malignant disease with propensity for systemic spread during the last 5 years
* Current or expected use of cytotoxic drugs
* Current untreated anaemia (e.g. sickle cell anaemia), i.e. Hb concentration < 11 g/dl (7 mmol/l)
* Use of recombinant erythopoetin
* Use of aprotinin and/or fibrin sealant
* Use of other autologous blood transfusion than that with the Sangvia® system (e.g. CellSaver, pre-donation, acute normovolemic haemodilution etc.)
* Women of childbearing age
* Fractures
* Revision/secondary total hip surgery with expected serious bone grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Poolman, Dr., Study Director — Onze Lieve Vrouwe Gasthuis (OLVG)
Locations (6):
- Medical University Vienna, Department of Orthopaedic Surgery, Vienna, Austria
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Reinier de Graaf Gasthuis (RdGG), afd. Orthopedie, Delft
  - MC Haaglanden, Orthopedic Dept., The Hague
- St. Olavs Hospital, Ortopedisk avdelning, Trondheim, Norway
- Hospital Universitario Mar- Esperança (IMAS), Servicio de Anestesiología, Barcelona, Spain

REFERENCES:
- [Derived] Thomassen BJ, Pilot P, Scholtes VA, Grohs JG, Holen K, Bisbe E, Poolman RW. Limit allogeneic blood use with routine re-use of patient's own blood: a prospective, randomized, controlled trial in total hip surgery. PLoS One. 2012;7(9):e44503. doi: 10.1371/journal.pone.0044503. Epub 2012 Sep 13. PMID 23028549

RESULTS

PARTICIPANT FLOW:
Groups:
- Sangvia: Autologous blood transfusion with Sangvia device (routinely)
- No Sangvia: No autologous blood transfusion.
Period: Overall Study
Arm/Group | Sangvia | No Sangvia
Started | 113 (7 participants excluded before surgery. No baseline data available) | 114 (4 participants excluded before surgery. No baseline data available)
Completed | 106 (APT/ITT analysis set) | 110 (APT/ITT analysis set)
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sangvia | No Sangvia | Total
Number analyzed (Participants) | 106 | 110 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 49 | 93
  >=65 years | 62 | 61 | 123
Age Continuous [Mean (Standard Deviation); unit: years] | 67 (11) | 65 (12) | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 70 | 146
  Male | 30 | 40 | 70
Region of Enrollment [Number; unit: participants]
  Spain | 5 | 5 | 10
  Austria | 12 | 13 | 25
  Norway | 7 | 6 | 13
  Netherlands | 82 | 86 | 168

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Need for Bank Blood Transfusion
Description: Bank blood transfusions were given in both groups after assessment of independent assessor, by using a transfusion trigger. All transfusions were recorded in a transfusion log and summarized at discharge. The total number of patients per group in need for any bank blood transfusion was compared.
  The participant were followed for the duration of hospital stay, an average of 6 days (SD 3 days)
Time Frame: At discharge
Population: Per protocol group. Major protocol deviations were excluded: Incorrect treatment, no treatment or exclusion criteria fulfilled.
Measure: Number; unit: Participants
Arm/Group | Sangvia | No Sangvia
Number analyzed (Participants) | 96 | 101
Participants | 9 | 13

ADVERSE EVENTS:
Arm/Group | Sangvia | No Sangvia
Serious Adverse Events (participants affected / at risk) | 7/106 | 7/110
Other Adverse Events (participants affected / at risk) | 12/106 | 9/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sangvia (N=106) | No Sangvia (N=110)
Cardiac insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hip dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infection hip (Infections and infestations) | 0 (0) | 1 (1)
Lung embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Luxation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Paralytic ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periprosthetic fissure (intra-operatively) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Saturation depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Suspected infection (positive bacterial culture) (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Wound leakage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sangvia (N=106) | No Sangvia (N=110)
Nausea (Gastrointestinal disorders) | 12 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days